CLINICAL TRIAL: NCT03394599
Title: Motivating Engagement for Physical Activity in the Elderly - Day Program
Brief Title: Motivating Videos to Encourage Cycling for Geriatric Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bruyère Health Research Institute. (Other)
Collaborators: Baycrest (Other); West Park Healthcare Centre (Other)
Responsible Party: Principal Investigator, Heidi Sveistrup, Interim CEO and Chief Scientific Officer of the Bruyère Research Institute and VP, Research and Academic Affairs, Bruyère Health Research Institute.
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Motiview Project
Record Dates: First submitted 2017-12-20; First posted 2018-01-09 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Physical Activity; Aging; Geriatrics
Keywords: Physical Activity; Rehabilitation; Exercise; Engagement; Older Adults
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TheraTrainer Only (Active Comparator): The 30 clients (15 per site) will have the opportunity to engage in cycling on the TheraTrainer only for the duration of their participation at the Geriatric program. Their carers will also be recruited.
  Interventions: Device: TheraTrainer Only
- TheraTrainer + Motiview (Experimental): The 30 clients (15 per site) will have the opportunity to engage in cycling on the TheraTrainer with the addition of Motiview (engaging videos to watching while cycling). Their carers will also be recruited.
  Interventions: Device: TheraTrainer + Motiview

INTERVENTIONS:
Device: TheraTrainer + Motiview — TheraTrainer will be used in conjunction with Motiview.
  Arms: TheraTrainer + Motiview
Device: TheraTrainer Only — TheraTrainer will be used.
  Arms: TheraTrainer Only

SUMMARY:
Motiview, an activity healthcare solution by Motitech, is finding solutions for elderly and people with dementia by reducing unnecessary emergency department visits, preventing falls/fall-injuries, improving management of complex health conditions, and improving brain health/cognitive fitness. Motiview is based on the premise that many of the challenges faced by this population may be caused by inactivity. The solution needs to effectively motivate them to be active year round. It also needs to accomplish this without increasing the resources within the health system. Motiview stimulates elderly people and people with dementia to increase their physical activity and cognitive training. By using videos, music/sound, the user can take a virtual bicycle trip through familiar surroundings and memories while facilitating activity participation and adherence in the older adult. Motiview is coupled to a mobile user-adapted cycle-trainer (TheraTrainer) that elicits physical activity as the individual pedals the trip. The unique part is adapting films and music according to the users' wishes and memories. By lessening the perceptions of difficulty, monotony, and discomforts associated with physical activity, participation and the experience of physical activity is enhanced. The research protocol of this project is designed to document the added value of Motiview for achieving physical activity participation. The hypothesis being that TheraTrainer bicycles will provide more activity when used with the video/audio overlay. Qualitative data will be gathered on the social aspects and reminiscence observed with the video/audit overlay from clients, care givers and staff.

Information about Motiview can also be found on the website at https://www.motitech.no/en

DETAILED DESCRIPTION:
Implementation will be conducted in two settings (Geriatric Day Hospital (GDH) Elisabeth Bruyere Hospital and the Day Treatment Centre (DTC) Baycrest Health Sciences). The settings selected have similar client profiles in terms of age, frailty, cognition, etc. Three subject groups will be included to obtain a holistic understanding of the use of this technology: geriatric program clients (clients) and their carers (carer) and staff (staff). All subjects (clients, carers and staff) will consent to participate prior to continuing with study involvement as documented below.

Recruitment and Consent:

- Baycrest -

Clients

DTC clients will undergo their usual intake assessment conducted by the DTC clinical team. Any clients who are determined to be medically unstable based on this assessment will not be recruited for this study. At the end of this assessment, any clients who are eligible for the study will be introduced to the study by the intake team. If they verbally consent to finding out more details about the project, their contact information will be provided to a research assistant (RA) who will then call the client with more information. If the client agrees to participate, they will be scheduled to meet the RA when they attend their regular DTC session during a time that does not conflict with treatment interventions or regular programming. At this point, the clients may choose to take part in a consenting session with the RA, followed by baseline testing. As a risk management strategy, the DTC clinical team will inform the research staff if a client is determined to be unable to continue participation at any point in the study.

Carers

Carers will be asked to contact the RA if they have any questions regarding the research project or if they would like to participate. On this call, the RA will confirm their understanding of their involvement in the research project. If the carers agree to participate, they will attend a session at Baycrest. During this session, the details of participation will be explained and the carers will be asked to repeat the information that has just been discussed, in order to ensure that they understand the consent form. Once they are fully informed, they will sign the consent form.

Staff

Following an informational session, consent forms will be left with the staff for them to read on their own. They will be told to contact the RA if they have any questions regarding the research project or if they decide to participate. The RA will then go to them at the DTC to collect the consent form and will ensure understanding of their participation at this time.

- Bruyere -

Clients

On the initial intake call by the GDH staff, all clients will be informed that there are research projects at the GDH that they may be eligible for. A verbal consent to contact will be obtained over the phone during this initial call. Contact information will then be sent to a recruitment coordinator who will then obtain consent for chart review to assess for eligibility for the research projects. Provided the client meets the inclusion criteria for the research project, the recruitment coordinator will then call back to inform them that they are eligible for participation and asked for verbal consent to be contacted by a member of the research team. If the client agrees to participate, they will be then invited to Bruyere prior to their GDH program to provide written consent and for baseline testing.

Carers

Following consenting and baseline testing with the client, the client will be told that the project is also interested in the perceptions of carers (family, informal carers). Clients will be asked to inform their carers of the study and to provide the RA's contact information so the carer can call with any questions. The carer will be subsequently invited to attend the baseline testing to provide written consent and to complete a semi-structured interview.

Staff

An informational session regarding Motiview will be provided to inform staff about the research project. Consent forms will be left at the end of the meeting for staff to read through on their own. If they decide to participate, they can leave their signed forms with the GDH reception for the research assistant in sealed envelopes that will be provided to them.

Study methods:

- Baycrest -

Clients

Participation: After the consenting and initial (baseline) testing session (which will be held at a time convenient to the client attending the DTC program, and which does not interfere with their regular programming/treatment intervention), the client will attend their day treatment program as usual (i.e., 3 hours a day, twice a week on either Monday & Wednesday or Tuesday & Thursday, for a duration of approximately 12 weeks). At Baycrest, assignment to the experimental or control group will be determined by their day treatment program schedule. If clients are scheduled for their program on Monday and Wednesday, they will be provided with the opportunity to use the TheraTrainer with Motiview (Experimental group). If they are scheduled for the program on Tuesday and Thursday, they will be provided with the opportunity to use the TheraTrainer without Motiview (allocated to the control group). Both groups will be informed that they have the option to use the TheraTrainer during any free time between their scheduled treatment appointments, for the duration of their day treatment program. Free time was selected so as to not disrupt a client's regularly scheduled treatment plans.

Every time a participant chooses to use the TheraTrainer, an occupational/physical therapy assistant hired for this project will assist the participant with his/her safe transfer onto and from the TheraTrainer. The assistant will set up the TheraTrainer (and Motiview system, if applicable). The assistant will record any field notes (i.e. reminiscence) that are relevant for the study. After the completion of a cycling session, participants will be asked micro-interview questions once per week to collect qualitative data about their cycling session. In addition, the participants will be continuously observed by the occupational/physical therapy assistant for the duration of each cycling session in the event that any participant experiences adverse responses to the physical activity. If any concerns arise related to the participants' ability to safely continue the cycling session, the session will be ended.

Follow-up outcomes: At the end of the study, participants will be asked to attend a post-participation session where they will participate in a post-participation semi-structured interview.

Carers

Participation: After consent is obtained, the carers will be taken through a semi-structured interview to gain feedback about their opinions about their study partner's involvement with the TheraTrainer and/or Motiview. Also, they will be asked about their general characteristics.

Follow-up: None for this group.

Staff

Participation: Following the study period, the staff will be taken through a semi-structured interview to gain feedback about their opinions about the client's involvement with the TheraTrainer and/or Motiview. Also, staff will be asked about their general characteristics.

Follow-up: None for this group.

- Bruyere -

Client

Participation: If the GDH client agrees to participate, they will be invited, along with their caregiver to Bruyere for one visit of approximately 30 minutes prior to their participation in the GDH. During this session, they will be told again of their involvement requirements for this study and signed written consent will be obtained. Subsequently, baseline outcome measure testing will be done.

They will then attend the rehabilitation program as usual and will be encouraged by the staff as part of their regular GDH program to use the TheraTrainer (one group with Motiview, one group without Motiview). At certain times throughout the study, when a participant uses the TheraTrainer as part of this investigation, study staff will take field notes to capture the clients'/residents' level of social engagement, and other behavioural or anecdotal findings that may emerge immediately prior to, during, or shortly after the exercise session.

To assess clients' experiences, they will be approached by study staff once a week (on different days throughout the week, depending on the client's schedule). The study staff will ask the clients if they would like to answer a few short questions related to their experience with the TheraTrainer (either with or without Motiview). Following their assent, the clients will be asked a maximum of four short questions related to their exercise experiences, reminiscence, and general health and well-being during each micro-interview. Each client will have the opportunity to take part in up to six micro-interviews in total throughout the study. The clients' responses will be audio recorded with their assent; for those who do not wish to have their responses recorded, study staff will take field notes related to the clients' responses instead (if assent is provided).

Follow-up: When each client has completed their GDH program, they will be asked to return to the Bruyere Continuing Care (room 441D) to complete the baseline outcome measures as a pre-post design.

Semi-structured interview questions will be posed to all clients who elect to take part in interview session as part of the study. The interviews will be held at the end of the study period. The questions and prompts were developed with the aim of employing a phenomenological approach, enabling the clients to elicit their own responses and experiences. Using the interview guide to lead the discussion, client responses may be probed to gain further clarity or insight. The interviews will be audio recorded by study staff. Study staff will also write field notes to document client responses and other observations to supplement and provide context for the transcripts.

Recruitment will continue until 15 clients (control group) have been enrolled and all have completed their geriatric rehabilitation program. After 15 clients have finished the study, Motiview will be placed into the GDH and recruitment of 15 (experimental group) additional clients will commence.

Carer

Same as Baycrest protocol.

Staff

Prior to the first client enrollment, staff will participate in a brief session (approximately 10 minutes) on proper use of the TheraTrainer, Motiview. The staff will be encouraged to use the TheraTrainer and Motiview as part of their rehabilitation protocol (TheraTrainer activity bikes will be used in place of the NuStep cycle currently in the GDH).

Semi-structured interview questions will be posed to all staff members who elect to take part in an interview session as part of the study. The interviews will be held after 15 clients use the TheraTrainer alone as well as after the 15 clients that use TheraTrainer and Motiview. The questions were developed with the aim of employing a phenomenological approach, which provides staff with the opportunity to elicit their own responses and experiences. Using the interview guide to lead the discussion, staff members' responses may be probed further to gain additional clarity or insight. The interviews will be audio recorded by study staff. Study staff will also write down field notes to capture any notable observations and to add further context to clients' responses, which will ultimately supplement the transcripts.

ELIGIBILITY:
Inclusion Criteria:

Clients-

* Will be attending the Geriatric Day Hospital program at Bruyere Continuing Care or the Day Treatment Centre at Baycrest Health Sciences
* Able to provide informed consent
* Able to safely use a TheraTrainer
* Would be using the exercise cycle as part of regular therapy in the GDH (Bruyere only) as determined by their health care team.

Carer-

* Able to provide informed consent.

Staff-

* Employed at the Geriatric Day Hospital/Day Treatment Centre program at the time of client enrollment.

Exclusion Criteria:

Client-

* Told by the therapists not to use the TheraTrainer as part of their rehabilitation.

Carer-

* No exclusion criteria

Staff-

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Psycho-social | Through study completion, an average of 8 weeks.
  Micro-interviews after use of the TheraTrainer

SECONDARY OUTCOMES:
Qualitative Feedback | One time, during the week following the intervention period.
  Post-intervention Semi-structured Interviews

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Sveistrup, PhD, Principal Investigator — Bruyère Health Research Institute.; Tim Pauley, MSc, Principal Investigator — West Park; Fidelma Serediuk, BSc PT, MSc, Principal Investigator — Baycrest
Locations (2):
- Canada (2):
  - Bruyere Research Institute, Ottawa, Ontario
  - Baycrest Health Sciences, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
All collected (de-identified) IPD will be shared between sites but not made accessible to other researchers.

DOCUMENTS (1):
  • Study Protocol (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/99/NCT03394599/Prot_000.pdf